CLINICAL TRIAL: NCT01554605
Title: Gait Disturbances and Hips Bone Mineral Density
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: TASMC-12-NV-648-CTIL
Record Dates: First submitted 2012-02-23; First posted 2012-03-15 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Difference in BMD Between Both Hips

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

SUMMARY:
The objective of this study is to investigate the role of gait disturbance as a cause for difference in Bone Mineral Density (BMD) between both hips. Each subject will undergo the following tests: Functional Mobility Testing, Gait analysis, Motion Analysis, Assessments for Balance and Gait and Cognitive assessments.

ELIGIBILITY:
Inclusion Criteria:

1. differeneces in hips in Bone Mineral Density test in one group.
2. Age 40-80.

Exclusion Criteria:

1. bone disease,
2. arthritis,
3. congenital skeletal malformations,
4. pregnancy,
5. neurological disease

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: subjects will be recruited from the bone clinic
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2012-03